CLINICAL TRIAL: NCT05087875
Title: Pilot Test of an mHealth Intervention for Reducing Alcohol Use Among Adolescent and Young Adult Cancer Survivors
Brief Title: Evaluating an mHealth Intervention for Reducing Alcohol Use Among Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolyn Lauckner (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Carolyn Lauckner, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67410; R21CA261844 (NIH)
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Alcohol Use
MeSH Terms: conditions — Neoplasms; Alcohol Drinking | interventions — Ethanol; Economics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAC: Tracking and Reducing Alcohol Consumption (Experimental): The TRAC intervention focuses on increasing motivation and building skills to reduce alcohol use and involves 4, 30-minute sessions with an interventionist done via video chat or phone.
  Participants will complete smartphone-based self-monitoring of alcohol use. Each morning, participants complete a mobile survey indicating if they drank the previous day and if so, how many drinks they had. Surveys will be programmed using REDcap and sent via a link in the reminder text message. Additionally, participants will be prompted each evening and asked to complete a breathalyzer reading using a mobile app to determine blood alcohol content (BAC). If safety concerns are identified (e.g., BAC ≥0.30; blackouts), the interventionist will refer the AYA to a licensed provider with expertise in substance use treatment.
  Interventions: Behavioral: TRAC: Tracking and Reducing Alcohol Consumption
- Control (Active Comparator): Participants in the control group will receive educational materials regarding alcohol consumption and its link to cancer . They will also participate in smartphone monitoring of alcohol use on the same schedule as participants in the intervention group. This will allow us to compare daily alcohol use data between the two conditions and evaluate the added component of weekly counseling in TRAC.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: TRAC: Tracking and Reducing Alcohol Consumption — The TRAC intervention focuses on increasing motivation and building skills for avoiding triggers and managing situations that encourage alcohol consumption. Participants set goals for reducing their drinking and learn strategies to help them achieve those goals. It requires four 30-minute sessions with a counselor using mobile phones.
  Arms: TRAC: Tracking and Reducing Alcohol Consumption
Other: No intervention — The comparison group will be evaluated based on daily self-monitoring data.
  Arms: Control

SUMMARY:
The objective of this study is to adapt and test the feasibility of a 4-week motivational interviewing mHealth intervention, Tracking and Reducing Alcohol Consumption (TRAC), to reduce alcohol use among adolescent and young adult (AYA) cancer survivors during post-treatment survivorship.

At the end of this study, the feasibility data gathered will inform a definitive randomized controlled trial of TRAC-AYA to test the efficacy of the adapted intervention.

DETAILED DESCRIPTION:
For this study, the investigators will adapt and pilot an existing mHealth intervention (TRAC) to reduce alcohol use among AYAs as part of a randomized controlled trial. TRAC includes weekly phone sessions with an interventionist and incorporates smartphones for daily self-monitoring of alcohol use. Upon enrollment, participants will be randomized into either the intervention (TRAC) arm or control (education and daily self-monitoring) arm.

Researchers will conduct the study in Kentucky, which leads the nation in cancer incidence and mortality, has a higher incidence of AYA cancers compared to other states, is 40% rural, and encompasses over 100 medically underserved areas. Participants will be recruited from the University of Kentucky Markey Cancer Center and its affiliate institutions.

Preliminary data used for this study were collected from a study (PI: Lauckner, K01AA02530) testing the TRAC intervention with people living with HIV/AIDS, which has shown promising preliminary results, with high feasibility, acceptability, and encouraging preliminary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer between age 15-39
* Currently age 18-39
* 3 months-15 years post-treatment
* Meets criteria for risky alcohol use
* Reside in United States

Exclusion Criteria:

* Severe psychopathology

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Lauckner, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TRAC: Tracking and Reducing Alcohol Consumption: The TRAC intervention focuses on increasing motivation and building skills to reduce alcohol use and involves 4, 30-minute sessions with an interventionist done via video chat or phone.
  Participants will complete smartphone-based self-monitoring of alcohol use. Each morning, participants complete a mobile survey indicating if they drank the previous day and if so, how many drinks they had. Surveys will be programmed using REDcap and sent via a link in the reminder text message. Additionally, participants will be prompted each evening and asked to complete a breathalyzer reading using a mobile app to determine blood alcohol content (BAC). If safety concerns are identified (e.g., BAC ≥0.30; blackouts), the interventionist will refer the AYA to a licensed provider with expertise in substance use treatment.
  TRAC: Tracking and Reducing Alcohol Consumption: The TRAC intervention focuses on increasing motivation and building skills for avoiding triggers and managing situations that encourage alcohol consumption. Participants set goals for reducing their drinking and learn strategies to help them achieve those goals. It requires four 30-minute sessions with a counselor using mobile phones.
Period: Overall Study
Arm/Group | TRAC: Tracking and Reducing Alcohol Consumption | Control
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRAC: Tracking and Reducing Alcohol Consumption | Control | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.79 (4.65) | 28.76 (6.35) | 29.73 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 17 | 20 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 16 | 18 | 34
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eligible Participants Enrolling in the Study
Description: The primary feasibility outcome is enrollment, with a goal of 60% of eligible AYAs approached enrolling in the study. A higher percentage of individuals who enroll in the study indicate the intervention is accessible to the target population.
Time Frame: 17 months
Population: Overall Number of Participants Analyzed represents the number of participants screened eligible to enroll.
Measure: Number; unit: percentage of eligible who enrolled
Groups:
- Screened Eligible Participants: Participants who completed the screening survey and were determined to be eligible to participate in the study.
Arm/Group | Screened Eligible Participants
Number analyzed (Participants) | 60
percentage of eligible who enrolled | 66.7

2. Secondary Outcome: Percent of Participants Completing Follow-up
Description: One of the secondary feasibility outcomes is retention, with a goal of 60% of study participants completing follow-up. A higher percentage of individuals completing follow-up indicates a greater degree of acceptability of the intervention.
Time Frame: 10 weeks
Measure: Number; unit: percentage completing follow-up
Arm/Group | TRAC: Tracking and Reducing Alcohol Consumption | Control
Number analyzed (Participants) | 19 | 21
percentage completing follow-up | 100 | 90.5

3. Secondary Outcome: Percent of Participants Completing Majority of Intervention Sessions
Description: One of the secondary feasibility outcomes is intervention adherence, with a goal of 70% of participants completing the majority (3/4 or 75%) of intervention sessions. Higher percentages indicate a greater degree of acceptability of the intervention. This outcome was only measured among the intervention group.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | TRAC: Tracking and Reducing Alcohol Consumption
Number analyzed (Participants) | 19
percentage of participants | 100

4. Secondary Outcome: Average Percent of Daily Monitoring Tasks Completed
Description: Monitoring adherence is measured by the average percentage of daily surveys and breathalyzers completed by participants.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: average percentage completed
Arm/Group | TRAC: Tracking and Reducing Alcohol Consumption | Control
Number analyzed (Participants) | 19 | 21
average percentage completed
  Daily survey adherence | 97.5 (4.9) | 93.5 (11.9)
  Daily breathalyzer adherence | 93.4 (12.3) | 84.7 (25.6)

5. Other Pre Specified Outcome: Daily Drinking
Description: This outcome will be measured using participants' self-reported alcohol use on a 4-item survey. This will assess whether any alcohol was consumed, the number of drinks, time since last drink, and plans to drink later in the day. Higher reports of daily drinking indicate greater consumption of alcohol.
Time Frame: Daily for 6 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Blood Alcohol Content
Description: This will be measured using the BACTrack Mobile Pro breathalyzer, with results being sent to the study team via mobile app. Higher blood alcohol content indicates greater consumption of alcohol.
Time Frame: Daily for 6 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Alcohol Use
Description: This will be measured using the PROMIS SF Alcohol 7a, which is a 7-item questionnaire used to assess alcohol use over the past 30 days.
  Raw scores can range from 7-35. All PROMIS measures can be converted to T-scores, in which the raw score is rescaled into a standardized score with a mean of 50 of standard deviation of 10. A higher T-score indicates more alcohol use in the past 30 days.
Time Frame: Measured at baseline, post-intervention (6 weeks), and one month post-intervention (10 weeks)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Overall Health
Description: This will be measured using the PROMIS-29 plus 2 v2.1, a 31 item scale which provides an overall profile of health with sub-scales (i.e., physical function, depression, anxiety, ability to participate in social roles/activities, sleep disturbance, fatigue, pain interference, pain intensity).
  All PROMIS measures can be converted to T-scores, in which the raw score is rescaled into a standardized score with a mean of 50 of standard deviation of 10. A higher T-score indicates more of the concept being measured, which scores calculated separately for each of the subscales.
Time Frame: Measured at baseline, post-intervention (6 weeks), and one month post-intervention (10 weeks)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Self-efficacy
Description: Self-efficacy will be measured using the PROMIS Self-efficacy SF 4a, a 4-item assessment of overall confidence in one's ability to solve problems and cope.
  Scores can range from 4-16. All PROMIS measures can be converted to T-scores, in which the raw score is rescaled into a standardized score with a mean of 50 of standard deviation of 10. A higher T-score indicates higher self-efficacy.
Time Frame: Measured at baseline, post-intervention (6 weeks), and one month post-intervention (10 weeks)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Personal Control Over Alcohol Use
Description: This outcome will be measured using the Personal Control Scale, which consists of 15 items and assesses personal control over drinking in the past 90 days (at baseline; past 60 days for post-intervention), and perceived control over one's current drinking. Scores can range from 0-60. Higher scores on this scale indicate participants' perceiving to have a greater degree of personal control over their drinking.
Time Frame: Measured at baseline, post-intervention (6 weeks), and one month post-intervention (10 weeks)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Alcohol Negative Consequences
Description: This outcome will be measured using the PROMIS SF Alcohol Use-Negative Consequences 7a, which is a 7-item scale that assesses perceived negative consequences of using alcohol in the past 30 days (e.g. unreliable, social problems, judgement).
  Raw scores can range from 7-45. All PROMIS measures can be converted to T-scores, in which the raw score is rescaled into a standardized score with a mean of 50 of standard deviation of 10. A higher T-score indicates a higher degree of perception of negative consequences surrounding alcohol use in the past 30 days.
Time Frame: Measured at baseline, post-intervention (6 weeks), and one month post-intervention (10 weeks)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Alcohol Positive Consequences
Description: The PROMIS adult Alcohol Use - Positive Consequences item bank assesses positive personal outcomes of alcohol use over the past 30 days. These items cover physical (e.g., improved sleep, increased sexual desire), mental (e.g., happiness, creativity, positive self-image), and social (e.g., comfort around others, ease in talking to others) consequences of drinking.
  Raw scores can range from 7-45. All PROMIS measures can be converted to T-scores, in which the raw score is rescaled into a standardized score with a mean of 50 of standard deviation of 10. A higher T-score indicates a higher degree of perception of positive consequences surrounding alcohol use in the past 30 days.
Time Frame: Measured at baseline, post-intervention (6 weeks), and one month post-intervention (10 weeks)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Tobacco Use
Description: This outcome will be measured using the Cancer Patient Tobacco Use Questionnaire (core items), which is a 4-item survey that assesses participants' lifetime and current tobacco use. This questionnaire is not scored.
Time Frame: Measured at baseline, post-intervention (6 weeks), and one month post-intervention (10 weeks)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Emotional Support
Description: Social support will be measured using the PROMIS Emotional Instrumental Support V2. This consists of 12 items, and assesses perceived emotional support and instrumental support (e.g. help with tasks).
  Raw scores can range from 12-60. All PROMIS measures can be converted to T-scores, in which the raw score is rescaled into a standardized score with a mean of 50 of standard deviation of 10. A higher T-score indicates a higher degree of emotional support.
Time Frame: Measured at baseline, post-intervention (6 weeks), and one month post-intervention (10 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment to end of study at 10 weeks.
Arm/Group | TRAC: Tracking and Reducing Alcohol Consumption | Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT05087875/Prot_SAP_ICF_001.pdf